CLINICAL TRIAL: NCT04182230
Title: UROGEN WEL-DONE: Can the Novel Rapid Diagnostic UROGEN WELL D-ONE Detect Common Causes of Urinary Tract Infections and Urethritis?
Brief Title: UROGEN WELL D-ONE : Evaluation of a Novel Diagnostic for Sexually Transmitted Bacterial Infections
Status: Completed | Type: Observational
Sponsor: Cwm Taf University Health Board (NHS) (Other Government)
Collaborators: Cardiff University (Other)
Responsible Party: Sponsor
Other Study IDs: CT 251053 3/07/18
Record Dates: First submitted 2019-11-27; First posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Sexually Transmitted Diseases, Bacterial; Bacterial Urinary Tract Infection; Antimicrobial Resistance
Keywords: Sexually transmitted infections
MeSH Terms: conditions — Sexually Transmitted Diseases, Bacterial; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention. This study was an evalution with no intervention. — Not an interventional study

SUMMARY:
UROGEN WELL D-ONE

Principal research question:

Can the UROGEN WELL D-ONE assay detect urinary tract infections and urethritis in clinical samples from patients attending Genitourinary Medicine outpatient clinics as accurately as standard laboratory microscopy and culture methodologies, while simultaneously identifying antimicrobial resistance?

The primary aim of this study is to evaluate the rapid diagnostic assay UROGEN WELL D-ONE and determine if it can accurately detect infectious organisms causing UTI's and urethritis.

Secondary research question:

Is the antimicrobial resistance identified by the UROGEN WELL D-ONE assay accurate as compared to determination by the Clinical and Laboratory Standards Institute international guidelines?

The secondary research objective will be to assess the accuracy of the breakpoint antimicrobial susceptibility measurement by the assay. This is particularly important with the global increase in antibiotic resistance, when the acquisition of mobile resistance genes to the remaining effective therapeutics is rising internationally.

DETAILED DESCRIPTION:
UROGEN WELL D-ONE is a new rapid culture-based benchtop diagnostic for the detection of urinary tract infections and urethritis. It detects the causative organisms and determines their antibiotic resistance. The novel test can detect bacterial infections such as E. coli, Staphylococcus spp., Enterococcus, Group B Streptococci, Mycoplasma spp, Ureaplasma spp, Neisseria spp, Gardnerella vaginalis, the protozoa Trichomonas vaginalis and Candida albicans. As such this diagnostic could be a very good tool to detect infection, identify the organism responsible for infection and with determination of antimicrobial susceptibility, guide treatment of these infections.

BACKGROUND- Urinary tract infections (UTIs) are a severe public health problem and are caused by a range of pathogens. High recurrence rates and increasing antimicrobial resistance among uropathogens threaten to greatly increase the economic burden of these infections. Urinary tract infections (UTIs) are some of the most common bacterial infections, affecting 150 million people each year worldwide1 UTIs are caused by both Gram-negative and Gram-positive bacteria, as well as by certain fungi. The most common causative agent for both uncomplicated and complicated UTIs is uropathogenic Escherichia coli (UPEC). For the agents involved in uncomplicated UTIs, UPEC is followed in prevalence by Staphylococcus saprophyticus, Enterococcus faecalis, group B Streptococcus (GBS), Neisseria spp., Staphylococcus aureus and Candida spp.2-5 Multidrug-resistant uropathogenic organisms are becoming an expanding public health threat, as Enterobacteriaceae family members increasingly acquire extended-spectrum β-lactamases, such as cefotaximases, oxacillinases, AmpC-type β-lactamases and carbapenemases.8-9. Routine testing techniques currently used for antibiotic sensitivity of pathogens causing UTIs can take 2-3 days to perform and so accurate treatment is often delayed. This delays treatment and can lead to increased morbidity.

Urethritis or inflammation of the urethra, is a multifactorial condition which is sexually acquired in the majority of (but not all) cases. It is characterised by urethral discharge, dysuria and/or urethral discomfort. Urethritis is described as either gonococcal, when Neisseria gonorrhoeae is detected, or nongonococcal (NGU) when it is not. Organisms implicated in this disease are commonly Chlamydia trachomatis, Mycoplasma spp, Ureaplasma spp, Trichomonas vaginalis and Candida. A number of studies indicate that antibiotic resistance in some of these organisms leads to microbiological failure of treatment, up to 68% for tetracyclines.11,13,14 , up to 33% for macrolides 10,11,13-18 and that mutations in the quinolone-resistance determining regions (QRDRs) of the gyrA and parC genes can occur with a prevalence of 10%19. Persistent NGU, when symptoms do not resolve following treatment, occurs in 15%-25% of patients following initial treatment of acute NGU. Recurrent NGU is empirically defined as the recurrence occurs in 10%-20% of patients.12,20 The aetiology of persistent NGU is probably multifactorial with a persistent infectious agent being identified in 50% of cases.11,12,20,21 Currently, testing for the detection of UTI and urethritis is expensive, requires highly trained laboratory staff and takes 48-72 hours. This delays treatment and can lead to increased morbidity. However, UROGEN WELL D-ONE is a new rapid culture-based clinical diagnostic assay, which will improve clinical provision for the detection of the cause of urinary tract infections and urethritis from urine samples e.g E. coli, Gardnerella vaginalis, Group B Streptococcus, Staphylococcus aureus, Neisseria spp., Enterococcus, E. Coli, Mycoplasma and Ureaplasma spp, the protozoa Trichomonas vaginalis and Candida albicans. It will also demonstrate their antimicrobial susceptibility. Importantly it uses the correct CLSI antibiotic threshold concentrations to determine antimicrobial resistance and does not require specialist equipment.

In summary, UROGEN WELL D-ONE has the potential to allow rapid detection of the common organisms that cause UTI and urethritis and guide antibiotic treatment, with a turnaround time of 18 hours. This has highly significant positive outcomes for patients and reduce empirical treatment of infection.

ELIGIBILITY:
Inclusion Criteria:

Participants must be sexually active. Participants will only be able to consent to this study if they have read and understood the Participant Information Sheet and been consented by a research nurse.

Exclusion Criteria:

Patients aged under 16 years. Patients who are victims of sexual assault Patients who are not sexually active Patients who are deemed unable to give informed consent.

Ages: 16 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Patients identifying as male, female and transgender.
Study Population: Participants who sexually active and attending a walk-in sexual health clinic for sexually transmitted infection testing and contraception provision.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
UROGEN WELL D-ONE PRIMARY OUTCOME | 365 days
  The primary aim of this study is to evaluate the rapid diagnostic assay UROGEN WELL D-ONE and determine the sensitivity and specificity of the assay for the detection of sexually transmitted bacterial infections.

SECONDARY OUTCOMES:
UROGEN WELL D-ONE SECONDARY OUTCOME | 365 days
  To determine the specificity and sensitivity of the assay for detection of antimicrobial resistance of bacteria and compare to determination by the Clinical and Laboratory Standards Institute international guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Lucy C Jones, DM, Principal Investigator — Cwm Taf University Health Board
Locations (1):
- Department of Sexual Health, Cwm Taf University Health board, Llantrisant, United Kingdom

IPD SHARING:
Plan to Share IPD: No